CLINICAL TRIAL: NCT03274414
Title: A Phase II, Single-Arm Trial Assessing Local Control of Near Total Endoscopic Resection Followed by Concurrent Chemotherapy and Proton Radiation in the Treatment of Unresectable Sinonasal Tumors
Brief Title: A Clinical Trial of Endoscopic Surgery Followed by Chemotherapy and Proton Radiation for the Treatment of Tumors in the Sinus and Nasal Passages
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-442
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2023-01

CONDITIONS: Paranasal Sinus Cancer; Nasal Cavity Tumor; Nasal Cavity Adenocarcinoma
Keywords: squamous cell carcinoma; esthesioneuroblastoma; adenoid cystic carcinoma; adenocarcinoma; cisplatin; 17-442
MeSH Terms: conditions — Paranasal Sinus Neoplasms; Carcinoma, Squamous Cell; Esthesioneuroblastoma, Olfactory; Carcinoma, Adenoid Cystic; Adenocarcinoma | interventions — Cisplatin; Endoscopic Mucosal Resection; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Unresectable paranasal sinus/nasal cavity malignancy (Experimental)
  Interventions: Drug: Cisplatin; Radiation: Adjuvant Proton Radiotherapy; Procedure: Endoscopic Resection; Drug: cisplatin and etoposide

INTERVENTIONS:
Drug: Cisplatin — Cisplatin should be administered on day 1 (+/- 3 days) of the start of radiotherapy and then every 3 weeks (unless there is a delay for safety concerns such as neutropenia) for a total of 3 cycles. 100 mg/m^2 (dose reductions after the first cycle allowed for toxicity)
Radiation: Adjuvant Proton Radiotherapy — Proton therapy treatment will follow the National Cancer Institute's "Guidelines for the Use of Proton Radiation Therapy in NCI-Sponsored Cooperative Group Trials". Proton therapy techniques may include passively scattered or scanning or pencil beam technology.
Procedure: Endoscopic Resection — In brief, an endoscope is used and two surgeons perform the intervention in a binostril manner. Tumor is generally resected with an emphasis on identification of the attachments in the paranasal sinuses, nasal cavity, or skull base.
Drug: cisplatin and etoposide — If the final surgical pathology report shows SNUC, at the discretion of the treating medical oncologist, the patient will receive an addition of etoposide chemotherapy to cisplatin chemotherapy. The dose of cisplatin will be decresed from 100 mg/m2 to 60 mg/m2. Cisplatin should be administered on days 1-2, 21-22 and 42-43 at a dose of 60 mg/m2 and Etoposide should be administered at days 1-3, 21-23, and 42-44 at a dose of 120 mg/m2.

SUMMARY:
This study is being done to test a new treatment plan for large tumors in the sinus or nasal cavity that will include endoscopic surgery plus chemotherapy and proton-beam radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years.
* Histopathologically confirmed diagnosis of one the following cancer types:

  * Squamous cell carcinoma
  * Esthesioneuroblastoma
  * Adenoid cystic carcinoma
  * Adenocarcinoma
* Paranasal sinus/nasal cavity malignancy is considered unresectable with negative margins surgery or resection would be considered excessively morbid. This could include lesions with:

  * Carotid involvement
  * Cavernous sinus invasion
  * Brain invasion
  * Orbital apex
  * Intraconal space
  * Pterygoid musculature involvement
  * Invasion of the clivus
* Resection of at least 80% of the volume of the tumor is feasible. Resectability will be determined by the surgeon and radiologist after discussion among the multidisciplinary team. For patients who have had surgery at an outside institution, the same parameters will be thoroughly screened to ensure the patient met the same inclusion criteria and resection standards.
* Patients must be a candidate for surgery (as per treating surgeon) and be able to tolerate proton radiation and chemotherapy (as per treating radiation oncologist and medical oncologist).
* Karnofsky performance statue >/= 70
* The subject has organ and marrow function and laboratory values rendering safe administration of Cisplatin:

  * The ANC >/= 1000/mm3 without colony stimulating factor support
  * Platelets >/= 100,000/mm3
  * Hemoglobin >/= 9 g/dL
  * Bilirubin </= 1.5 mg/dL the ULM. For subjects with Gilbert's disease, bilirubin </= 3.0 mg/dL
  * Serum albumin >/= 2.8 g/dl
  * Creatinine clearance (CrCl) >/= 60 mL/min. For creatinine clearance estimation, the Cockcroft and Gault equation should be used:
  * Male: CrCl (mL/min) = (140 = age) x wt (kg) / (serum creatinine x 72)
  * Female: Multiply above result by 0.85
  * ALT and AST </= 3.0 ULN
  * Serum phosphorus, calcium, magnesium and potassium >/= LLN
* No evidence of intercurrent infection
* Negative pregnancy test for women of childbearing potential (<51 years of age) as per institutional policy.
* Patients with distant metastatic disease may not be included.
* Patient must be able to read and write in English.
* Patients who intitially meet the histopathological inclusion criteria but surgical pathology report shows Sinonasal Undifferentiated Carcinoma.

Exclusion Criteria:

* Tumor is deemed to be resectable with negative margins by conventional surgical standards.
* Patients not able to receive standard-dose cisplatin based on the judgement of the treating medical oncologist.
* Patients with chronic kidney disease (GFR <60), uncontrolled hypertension, congestive heart failure, pre-existing bone marrow dysfunction, or cytopenias.

  ° Congestive heart failure (CHF): New York Heart Association (NYHA) Class II-IV at the time of screening
* Concurrent uncontrolled hypertension defined as sustained blood pressure > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment; If severe hearing impairment is measured or if significant neuropathy is reported at baseline the treating physician will discuss the risks for further permanent hearing loss and neuropathy with the patient.
* Patients not able to have a MRI (due to pacemaker, claustrophobia, etc.).
* Inability to return to MSKCC for frequent scheduled hydration sessions post-chemotherapy.
* Inability to comply with requirements for cisplatin administration anti-emetic regimens post-treatment.
* Patients not able or unwilling to travel for proton therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Cohen, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memoral Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memoral Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Unresectable Paranasal Sinus/Nasal Cavity Malignancy: cisplatin and etoposide
Period: Overall Study
Arm/Group | Unresectable Paranasal Sinus/Nasal Cavity Malignancy
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Unresectable Paranasal Sinus/Nasal Cavity Malignancy
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 60 [38 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Local Control Assessment of Unresectable Paranasal Sinus and Nasal Cavity Tumors
Description: Assessment of local control after near-total endoscopic resection (NTR) followed by concurrent chemotherapy with proton-beam radiation in unresectable tumors (which we define as expected inability to perform negative margin surgery) of the paranasal sinuses and nasal cavity.
Time Frame: 1 year
Population: N/A - data were not collected
Arm/Group | Unresectable Paranasal Sinus/Nasal Cavity Malignancy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Unresectable Paranasal Sinus/Nasal Cavity Malignancy
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT03274414/Prot_SAP_000.pdf